CLINICAL TRIAL: NCT00986752
Title: Randomized Trial of Stenting After Dilation With or Without Paclitaxel Eluting Balloon or Atherectomy in Patients With Symptomatic Peripheral Artery Disease
Brief Title: Efficacy Study of Stenting, Paclitaxel Eluting Balloon or Atherectomy to Treat Peripheral Artery Disease
Acronym: ISAR-STATH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GE IDE No. B00101
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2010-01

CONDITIONS: Peripheral Vascular Diseases
Keywords: stent; atherectomy; paclitaxel-eluting balloon
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Stents; Atherectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stenting (Active Comparator): Due to randomization one nitinol stent will be implanted after dilation with a conventional balloon.
  Interventions: Device: Stenting (Smart Stent)
- Stenting after PEB (Experimental): Due to randomization one nitinol stent will be implanted after dilation with a Paclitaxel eluting balloon.
  Interventions: Device: Stenting (Smart Stent); Device: Stenting after PEB (Smart Stent, Invatec)
- Atherectomy (Experimental): The third randomization arm is Atherectomy.
  Interventions: Procedure: Atherectomy (SilverHawk device)

INTERVENTIONS:
Device: Stenting (Smart Stent) — Nitinol stent
  Other Names: Smart Stent, Cordis, Johnson & Johnson
  Arms: Stenting; Stenting after PEB
Device: Stenting after PEB (Smart Stent, Invatec) — Stenting (nitinol stent) after dilation with Paclitaxel-eluting balloon (PEB).
  Other Names: Invatec; Smart Stent, Cordis, Johnson & Johnson
  Arms: Stenting after PEB
Procedure: Atherectomy (SilverHawk device) — Atherectomy
  Other Names: SilverHawk device (EV3 Inc)
  Arms: Atherectomy

SUMMARY:
The purpose of the study is to evaluate the efficacy of stenting after dilation with or without paclitaxel-eluting balloon or atherectomy in patients with symptomatic peripheral artery disease.

DETAILED DESCRIPTION:
The superficial femoral artery is a common place for arteriosclerosis in patients symptomatic for lower extremity vascular disease. Advances in percutaneous transluminal angioplasty (PTA) and stenting have provided new options for the treatment of the disease in this arterial segment. Despite the initial technical success rate of more than 95% the late clinical failure remains an important concern.

Restenosis after PTA occurs in 40-60% within one year. Percutaneous removal of the obstructive material through atherectomy may reduce restenosis rate. So far, data in support of excisional atherectomy derive from registries. Another attempt to reduce restenosis is the use of paclitaxel eluting balloons (PEB). First clinical studies suggest that the use of PEBs during percutaneous treatment of femoropopliteal disease is associated with significant reductions in late lumen loss and target-lesion revascularization.

There is no randomized comparison of this three different interventional strategies. Thus the aim of this study is to evaluate the efficacy of these strategies in terms or reduction of diameter stenosis at follow-up angiogram.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic ≥ 70% stenosis of the SFA (Rutherford stage 2-6)
* Written informed consent

Exclusion Criteria:

* Acute ischemia and/or acute thrombosis of the SFA
* Untreated ipsilateral iliac artery stenosis >70%
* Previous stenting of the SFA
* Popliteal stenosis >70%
* Severe renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Percentage diameter stenosis | 6 months

SECONDARY OUTCOMES:
All-cause mortality | 6 and 24 months
Major adverse peripheral events (MAPE) defined as acute thrombosis of SFA or ipsilateral amputation or revascularization (PTA or bypass surgery) | 6 months
Time to onset of any of MAPE. | 3-24 months
Binary restenosis rate | 6 months
Percentage diameter stenosis in duplex ultrasound | 6 and 24 months
Change from baseline in functional status and health related quality of life (Walking Impairment Questionaire) | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, MD, Study Chair — Deutsches Herzzentrum München; Ilka Ott, MD, Principal Investigator — Klinikum rechts der Isar
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum, München
  - I. Medizinische Klinik, Klinikum rechts der Isar, München

REFERENCES:
- [Derived] Ott I, Cassese S, Groha P, Steppich B, Hadamitzky M, Ibrahim T, Kufner S, Dewitz K, Hiendlmayer R, Laugwitz KL, Schunkert H, Kastrati A, Fusaro M. Randomized Comparison of Paclitaxel-Eluting Balloon and Stenting Versus Plain Balloon Plus Stenting Versus Directional Atherectomy for Femoral Artery Disease (ISAR-STATH). Circulation. 2017 Jun 6;135(23):2218-2226. doi: 10.1161/CIRCULATIONAHA.116.025329. Epub 2017 Apr 19. PMID 28424222